CLINICAL TRIAL: NCT06275620
Title: A Phase 1/2 Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of AGTC-501 (rAAV2tYF-GRK1-RPGR) and a Phase 2 Randomized, Controlled, Masked, Multi-center Study Comparing Two Doses of AGTC-501 in Male Participants With X-linked Retinitis Pigmentosa
Brief Title: A Study Comparing Two Doses of AGTC-501 in Male Participants With X-linked Retinitis Pigmentosa Caused by RPGR Mutations (DAWN)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGTC-RPGR-001 DAWN
Record Dates: First submitted 2024-02-16; First posted 2024-02-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; retinal degeneration; RPGR; adeno-associated virus; gene therapy; AAV
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (High Dose, Standard Corticosteroid) (Experimental): Following a pars plana vitrectomy, the previously untreated eye of participants (n=up to 12) will receive a central subretinal injection at the high dose in the study eye at the Baseline visit; no treatment will be administered in the previously treated fellow eye.
  The corticosteroid taper for all treated participants in Groups 1 and 2 (high and low doses with standard corticosteroid regimen) will be a standard taper over the course of several weeks.
  Interventions: Biological: AGTC-501 (high dose and standard corticosteroid regimen)
- Group 2 (Low Dose, Standard Corticosteroid) (Experimental): Following a pars plana vitrectomy, the previously untreated eye of participants (n=6) will receive a central subretinal injection at the low dose in the study eye at the Baseline visit; no treatment will be administered in the previously treated fellow eye.
  The corticosteroid taper for all treated participants in Groups 1 and 2 (high and low doses with standard corticosteroid regimen) will be a standard taper over the course of several weeks.
  Interventions: Biological: AGTC-501 (low dose and standard corticosteroid regimen)
- Group 3 (High Dose, Modified Corticosteroid) (Experimental): Following a pars plana vitrectomy, the previously untreated eye of participants (n=approximately 3-6) will receive a central subretinal injection at the high dose in the study eye at the Baseline visit; no treatment will be administered in the previously treated fellow eye.
  Participants in Group 3 (high dose, modified corticosteroid) will have a more rapid corticosteroid taper.
  Interventions: Biological: AGTC-501 (high dose and modified corticosteroid regimen)

INTERVENTIONS:
Biological: AGTC-501 (high dose and standard corticosteroid regimen) — Adeno-associated virus vector expressing a human RPGR gene
  Arms: Group 1 (High Dose, Standard Corticosteroid)
Biological: AGTC-501 (low dose and standard corticosteroid regimen) — Adeno-associated virus vector expressing a human RPGR gene
  Arms: Group 2 (Low Dose, Standard Corticosteroid)
Biological: AGTC-501 (high dose and modified corticosteroid regimen) — Adeno-associated virus vector expressing a human RPGR gene
  Arms: Group 3 (High Dose, Modified Corticosteroid)

SUMMARY:
This Phase 2 study is a non-randomized, open-label, study of the safety of AGTC-501 in participants with XLRP who have previously been treated with a full-length AAV vector-based gene therapy targeting RPGR protein.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, multicenter study to evaluate the safety of 2 doses of AGTC-501 administered as a single subretinal injection in participants with XLRP who have previously been treated with a full-length AAV vector-based gene therapy targeting RPGR protein.

The trial includes a screening period of up to 60 days and a 5 year study period.

Each participant will receive a single subretinal injection of one of two dose levels of AGTC-501 in their previously untreated eye. There will be 3 groups. Group 1 will receive the high dose and include up to 12 participants, Group 2 will receive the low dose and will include 6 participants, and Group 3 will include ~3-6 participants. Participants in Groups 1 and 2 will receive the standard corticosteroid regimen. A single subretinal injection of the high dose AGTC-501 will be administered to participants in Group 1 (n = 12), while participants in Group 2 (n = 6) will receive a single subretinal injection of low dose AGTC-501. Group 2 (low dose AGTC-501, Standard Steroid) will be dosed before moving to Group 3. After 6 Group 1 (high dose) study participants reach post-operative Month 1, all data will be reviewed by the DSMC. If no safety signals arise, additional participants, Group 3 (n ~ 3-6), will receive a single subretinal injection of the high dose with a modified course of corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥12 years of age
* Have one eye previously treated with an AAV vector-based gene therapy designed to provide full-length functioning RPGR protein.
* Have a BCVA no better than 78 letters and no worse than 34 letters
* Be able to perform all tests of visual and retinal function and structure in both eyes based on the participant's reliability and fixation, per the Investigator's discretion.
* Have detectable baseline mean macular sensitivity measured by MAIA microperimetry, as determined by the Investigator and confirmed by the Central Reading Center (CRC).
* Have detectable EZ line in the study eye as assessed by SD-OCT and confirmed by the CRC.

Exclusion Criteria:

* Have other known disease-causing mutations documented in the participant's medical history or identified through a retinal dystrophy gene panel that, in the opinion of the Investigator, would interfere with the potential therapeutic effect of the study agent or the quality of the assessments.
* Have pre-existing eye conditions that would preclude the planned surgery, interfere with the interpretation of study endpoints, or increase the risk of surgical complications
* Had intraocular surgery within 90 days of study treatment administration.
* Have any active ocular/intraocular infection or inflammation
* Have a history of steroid-induced raised IOP of >25 mmHg following corticosteroid exposure, despite topical IOP-lowering pharmacologic therapy.

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The primary safety outcome is the number of participants experiencing Grade 3 or higher local (ocular) or non-ocular treatment-emergent adverse events, including treatment-emergent serious adverse events (SAEs). | Day 0 - Month 12
The primary safety outcome is the proportion of participants experiencing Grade 3 or higher local (ocular) or non-ocular treatment-emergent adverse events, including treatment-emergent serious adverse events (SAEs). | Day 0 - Month 12

SECONDARY OUTCOMES:
The number of participants experiencing treatment-emergent AEs of ocular/non-ocular adverse events, including treatment-emergent serious AEs. | Day 0 - Month 12
The proportion of participants experiencing treatment-emergent AEs of ocular/non-ocular adverse events, including treatment-emergent serious AEs. | Day 0 - Month 12
Change from baseline in mean sensitivity across the whole grid, as measured by MAIA (Macular Integrity Assessment) microperimetry, assess photoreceptor function under low light | Day 0 - Month 12
Response, as measured by MAIA (Macular Integrity Assessment) microperimetry, where response is defined as a greater than or equal to 7 decibel (dB) visual sensitivity improvement from baseline in at least 5 loci. | Day 0 - Month 12
Change from baseline in full-field stimulus threshold (FST) | Day 0 - Month 12
  As assessed by full-field stimulus threshold (FST); FST measures the sensitivity of the visual field by testing for the lowest luminance flash which elicits a visual sensation perceived
Change from baseline in Best Corrected Visual Acuity (BCVA) using Early-Treatment Diabetic Retinopathy Study (ETDRS) visual acuity | Day 0 - Month 12
Change from baseline in Low Luminance Visual Acuity (LLVA) using Early-Treatment Diabetic Retinopathy Study (ETDRS) visual acuity | Day 0 - Month 12
Proportion of responding eyes in treated versus control eyes at Month 12 where responder is defined as an improvement of at least 15-letters on low-luminance visual acuity (LLVA) | Day 0 - Month 12
Change from baseline in ellipsoid zone (EZ) area measured by spectral domain optical coherence tomography (SD OCT) | Day 0 - Month 12
Change from baseline in seven domain scores from a Michigan Retinal Degeneration Questionnaire (MRDQ) | Day 0 - Month 12
Change from baseline in Ora-VNC (visual navigation course) mobility test score | Day 0 - Month 12
  As assessed by functional assessment Ora-VNC (visual navigation course) mobility course
Change from baseline in the MObility Standardized Test-Virtual Reality (MOST-VR) mobility course test score | Day 0 - Month 12
  As measured by the MObility Standardized Test-Virtual Reality (MOST-VR) mobility course

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Florida, Jacksonville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Boston Children's Hospital, Boston, Massachusetts
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876